CLINICAL TRIAL: NCT01615731
Title: Value of Mifepristone in Eliminating the Need for a Second Set of Osmotic Dilators Prior to Dilation and Evacuation Between 19-24 Weeks: A Randomized Trial
Brief Title: Value of Mifepristone in Cervical Preparation Prior to Dilation and Evacuation 19-24 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-05302012-10088
Record Dates: First submitted 2012-05-30; First posted 2012-06-11 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Abortion, Induced
Keywords: Mifepristone; Induced Abortion; Dilation and Evacuation; Cervical preparation; Osmotic dilators
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two sets of dilators (Active Comparator): Two sets of osmotic dilators inserted 1 and 2 days pre-op
  Interventions: Other: Hygroscopic cervical dilators; Drug: Misoprostol; Drug: Intra-amniotic digoxin
- Mifepristone plus one set of dilators (Experimental): One set of dilators plus mifepristone
  Interventions: Drug: Mifepristone; Other: Hygroscopic cervical dilators; Drug: Misoprostol; Drug: Intra-amniotic digoxin

INTERVENTIONS:
Drug: Mifepristone — 200mg Mifepristone orally
  Other Names: Danco, Mifeprex
  Arms: Mifepristone plus one set of dilators
Other: Hygroscopic cervical dilators — Dilapan-S osmostic cervical dilators inserted through the internal os
  Other Names: Dilapan-S
Drug: Misoprostol — 400mcg buccal misoprostol 90 minutes pre-op
Drug: Intra-amniotic digoxin — 1mg digoxin administered intra-amniotically ~24 hours pre-op

SUMMARY:
A common practice for preparation for surgical abortion after 19 weeks gestation is the placement of multiple sets of osmostic dilators 1-2 days prior to the procedure. The investigators aim to study the addition of mifepristone as an adjunct to cervical dilation prior to abortion between 19-24 weeks gestation, and its potential to minimize the number of painful procedures and time in clinic (or away from work/home) that multiple sets of dilators can require. The investigators hypothesize that one set of dilators with mifepristone will result in similar procedure times and decreased "total" time as two sets of dilators.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Viable, Singleton pregnancy
* Voluntarily seeking abortion between 19 and 24wks gestation
* Able to give informed consent and comply with study protocol
* Fluent in English or Spanish

Exclusion Criteria:

* Allergy to misoprostol or mifepristone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University Medical Center, Stanford, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Started | 24 | 26
Completed | 21 | 24
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (6.5) | 27.7 (6.7) | 27.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Measured as time from speculum insertion to removal
Time Frame: Intraoperative Time
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
minutes | 10.9 (5.1) | 11.8 (5.4)

2. Primary Outcome: Total Procedure Time
Time Frame: Measured at clinic visits and on OR day, over a 3 day period
Population: Data missing for two subjects in "Mifepristone plus one set of dilators" arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 22
hours | 165 (57) | 86 (44)

3. Secondary Outcome: Maximum Cervical Dilation
Description: Measured by estimate with bimanual exam and passage of largest dilator immediately prior to procedure.
Time Frame: Measured intra-operatively
Population: Data missing for one subject in "Mifepristone plus one set of dilators" arm.
Measure: Number; unit: participants
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 23
participants
  Pre-op Cervical Dilation 2 cm | 2 | 3
  Pre-op Cervical Dilation 3 cm | 9 | 14
  Pre-Op Cervical Dilation 4 cm | 8 | 5
  Pre-Op Cervical Dilation 5 cm | 2 | 1

4. Secondary Outcome: Adverse Events (EBL)
Description: One adverse event: Estimated Blood Loss
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
mL | 57 (31) | 63 (43)

5. Secondary Outcome: Ease of Procedure by Blinded Surgeon
Description: Used a Visual Analogue Scale to determine the ease of procedure by blinded surgeon. The VAS ranges from 0-100. 0 being the easiest procedure the surgeon felt they had every performed and 100 being the most difficult procedure imaginable by the surgeon.
Time Frame: Measured Immediately after procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
units on a scale | 29 [23 to 52] | 30 [18 to 49]

6. Secondary Outcome: Pain Perceived by Patient
Description: Used a Visual Analogue Scale to determine the pain perceived by the patient pre-operatively (after misoprostol, immediately before transport to OR) and post-operatively (in recovery room, on average 1.5 hours post-operatively). The VAS ranges from 0-100. 0 being no pain felt by the patient and 100 being the worst pain imaginable felt by the patient.
Time Frame: Measured pre-operatively (after misoprostol, immediately before transport to OR) and post-operatively (in recovery room, on average 1.5 hours post-operatively)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
units on a scale
  Subject Pain Pre-Op | 13 [7 to 34] | 63 [16 to 78]
  Subject Pain Post-Op | 3 [1 to 32] | 16 [6 to 29]

7. Secondary Outcome: Overall Patient Experience
Description: Used a Visual Analogue Scale to determine the patient's overall satisfaction with her experience. The VAS ranges from 0-100. 0 being a worse than expected experience, 50 being what the patient expected and 100 being a better than expected experience.
Time Frame: Measured post operatively (at least 30 minutes, on average 1.5 hours) prior to discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
units on a scale | 72 [66 to 91] | 79 [67 to 88]

8. Secondary Outcome: Adverse Events
Description: uterine perforation, uterine injury, etc.
Time Frame: Intraoperatively and 2 weeks post operatively
Measure: Number; unit: participants
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Number analyzed (Participants) | 21 | 24
participants
  Pre-Procedure Delivery | 2 | 1
  Cervical Injury | 0 | 1
  RUpture of Membranes with Subsequent Fever | 1 | 0

ADVERSE EVENTS:
Arm/Group | Two Sets of Dilators | Mifepristone Plus One Set of Dilators
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 3/24 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Two Sets of Dilators (N=24) | Mifepristone Plus One Set of Dilators (N=26)
Pre-Procedure Delivery (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Cervical Injury (Injury, poisoning and procedural complications) | 0 | 1
Rupture of Membranes with Subsequent Fever (Pregnancy, puerperium and perinatal conditions) | 1 | 0

LIMITATIONS AND CAVEATS:
Failure of randomization with respect to assigning similar numbers of nulliparous women to both groups; inaccurate method for measurement of pre-operative cervical dilation; small size of cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No